CLINICAL TRIAL: NCT05938413
Title: Community Health Worker And MHealth to ImProve Viral Suppression (CHAMPS Pilot)
Acronym: CHAMPS Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion (in Nursing) and Professor of Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU2064
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: HIV/AIDS
Keywords: ART; PLWH; HIV Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention or CHAMPS (Experimental): Wise App that delivers medication adherence reminders and community health worker sessions
  Interventions: Device: Wise App with medication adherence reminders; Behavioral: CHW Sessions
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: Wise App with medication adherence reminders — The Intervention group will receive the Wise App that delivers medication adherence reminders.
  Arms: Intervention or CHAMPS
Behavioral: CHW Sessions — The Intervention group will complete sessions with a community health worker (CHW).
  Arms: Intervention or CHAMPS

SUMMARY:
The overall goal of this study is to evaluate the feasibility of a remotely delivered CHAMPS intervention for people living with HIV (PLWH) in a randomized controlled trial. The proposed trial is scientifically significant in representing a principled and systematic effort to test the efficacy of a combined community health worker (CHW) and smartphone intervention linked to a smart pill box for antiretroviral (ART) adherence in PLWH in the United States (US). Guided by a rigorous theoretical model of supportive accountability and building on preliminary work, this intervention has the potential to enable PLWH to self-manage their ART regimens while CHW monitor their ART adherence in real-time ultimately leading to viral suppression and ART adherence.

DETAILED DESCRIPTION:
Persons living with HIV (PLWH) now achieve a near-normal life expectancy due to antiretroviral therapy (ART) which has transformed HIV from a terminal diagnosis to a manageable chronic condition. Despite widespread availability of ART in the United States (US), many of the country's approximate 1.1 million PLWH are not fully benefitting from ART due to poor adherence. These suboptimal HIV health outcomes occur at a time when clinicians have limited time and the US healthcare system remains fragmented, further exacerbating the challenges inherent in the lives of underserved, marginalized groups, such as PLWH. Therefore, the development and evaluation of interventions using a cadre of community health workers (CHW) holds promise for addressing these challenges in the US. This study addresses limitations in current research on CHW interventions to improve viral suppression and ART adherence. The ubiquitous nature of mHealth technologies in daily life creates opportunities for health behavior management tools that were not previously possible and has the potential to address many of the healthcare needs of PLWH. The investigators propose to build on strong preliminary data to strengthen a community health worker (CHW) intervention using an existing mHealth approach, and provide further information regarding the successful wide-scale implementation of this combination intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Able to speak, read, and write in English or Spanish;
2. Aged ≥18 years;
3. Willing to provide a valid form of identification for verification;
4. Willing to participate in any assigned arm of the intervention;
5. Having been diagnosed with HIV ≥6 months ago;
6. Have an HIV-1 RNA level >200 copies/mL as verified by provision of medical records, or have a detectable load of >500 copies/mL, as measured by dried blood spot (DBS) sample kits, or report either not being virally suppressed in the past 12 months or being virally unsuppressed in the past 12 months;
7. Own a smartphone;
8. Ability and willingness to provide informed consent for study participation and consent for access to medical records; and
9. Live in the United States

Exclusion Criteria:

1. Reside in a nursing home, prison, and/or receiving in-patient psychiatric care at time of enrollment;
2. Terminal illness with life expectancy <3 months;
3. Planning to move out of the country in the next 3months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, RN, Principal Investigator — Columbia University School of Nursing
Locations (1):
- Columbia University School of Nursing, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shourya S, Liu J, McInerney S, Casimir T, Kenniff J, Kershaw T, Batey D, Schnall R. A Remote Intervention Based on mHealth and Community Health Workers for Antiretroviral Therapy Adherence in People With HIV: Pilot Randomized Controlled Trial. JMIR Form Res. 2025 Apr 2;9:e67997. doi: 10.2196/67997. PMID 40173448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention or CHAMPS
Started | 20 | 20
Completed | 18 | 12
Not Completed | 2 | 8
Not completed — Lost to Follow-up | 1 | 7
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention or CHAMPS | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (13.52) | 46.5 (11.89) | 47.85 (12.64)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 12 | 24
  Female | 7 | 8 | 15
  Something Else | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 9 | 5 | 14
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Relationship Status [Count of Participants; unit: Participants]
  Single | 10 | 14 | 24
  In a relationship with a man | 6 | 3 | 9
  In a relationship with a woman | 1 | 0 | 1
  Divorced/separated from a man | 1 | 0 | 1
  Divorced/separated from a woman | 1 | 0 | 1
  Widowed | 0 | 1 | 1
  Other | 1 | 2 | 3
Children [Count of Participants; unit: Participants] — Are a parent to a child or children.
  Participants
    No | 12 | 15 | 27
    Yes | 8 | 5 | 13
Highest Level of Education [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Elementary School | 0 | 0 | 0
  Some high school, no diploma | 2 | 3 | 5
  High school diploma or equivalent | 5 | 5 | 10
  Some college | 6 | 4 | 10
  Associate degree or technical degree | 4 | 3 | 7
  Bachelor/college degree | 2 | 3 | 5
  Professional or graduate degree | 1 | 2 | 3
Viral Load [Count of Participants; unit: Participants] — Using dried blood spot samples or electronic health records obtained during study visits, viral load levels will be used to assess ART adherence. The number of participants with detectable viral load (>=200 copies/mL in electronic health record (EHR), >=500 copies/mL in DBS) and not detectable viral load (<200 copies/mL in EHR, <500 in dried blood spot (DBS)) will be reported.
  Participants
    Viral Load Not Detectable | 17 | 11 | 28
    Viral Load Detectable | 3 | 9 | 12
Score on the Self-Rating Scale Item [Mean (Standard Deviation); unit: units on a scale] — The Self-Rating Scale Item is a single-item self-report adherence measure that uses a 6-point Likert scale to describe medication adherence over the past 4 weeks. Scores range from 1(very poor) to 6 (excellent).
  units on a scale | 4.80 (1.34) | 4.9 (1.35) | 4.85 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Viral Load
Description: Using dried blood samples or electronic health records obtained during study visits, viral load levels will be used to assess ART adherence. The number of participants with detectable viral load (>= 200 copies/mL in EHR; >= 500 copies/mL in DBS) and not detectable viral load (<200 copies/mL in EHR, <500 copies/mL in DBS) will be reported. The intervention effect at the 3 month follow up was adjusted for various values of baseline.
Time Frame: 3 months
Population: 17 analyzed as an insufficient sample was provided by n=1 (did not yield a result)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention or CHAMPS
Number analyzed (Participants) | 17 | 12
Participants
  Viral Load Not Detectable | 15 | 11
  Viral Load Detectable | 2 | 1
Statistical Analysis 1: Comparison: Control vs Intervention or CHAMPS; Test type: Non-Inferiority — Non-inferiority test to compare viral suppression rate between month 3 and baseline; Odds Ratio (OR) = 3.01

2. Secondary Outcome: Antiretroviral Therapy (ART) Adherence - CleverCap
Description: The CleverCapTM dispenser will automatically record each time a participant opens the dispenser. The investigators will collect adherence data each day from the start to the end of trial (day 1 to 3 months), and it is a count response (number of times taking medication each day). The percentage of their prescribed doses taken will be reported.
Time Frame: Up to 3 months
Population: This outcome measures ART adherence using CleverCap. The control group is not reported in this outcome as they were not exposed to the intervention and therefore did not receive the CleverCap device.
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses
Arm/Group | Intervention or CHAMPS
Number analyzed (Participants) | 12
percentage of prescribed doses | 60.08 (19.15)

3. Secondary Outcome: Score on the Self-Rating Scale Item (SRSI)
Description: The Self-Rating Scale Item is a single-item self-report adherence measure that uses a 6-point Likert scale to describe medication adherence over the past 4 weeks. Scores range from 1(very poor) to 6 (excellent).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention or CHAMPS
Number analyzed (Participants) | 18 | 12
score on a scale | 5.27 (1.23) | 5.25 (1.17)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control | Intervention or CHAMPS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05938413/Prot_SAP_000.pdf